CLINICAL TRIAL: NCT01805388
Title: Comparison of Tissue Formation in Regenerative Endodontic Procedures and Apexification
Brief Title: Comparison of Tissue in Regenerative Endodontic Procedures and Apexification
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of pediatric recruitment ability
Sponsor: Kenneth Hargreaves (Other)
Responsible Party: Sponsor-Investigator, Kenneth Hargreaves, Sponsor-Investigator, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC20130054H
Record Dates: First submitted 2013-02-28; First posted 2013-03-06 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Dental Pulp Regeneration
Keywords: Dental Pulp Regeneration
MeSH Terms: interventions — Root Canal Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regeneration Treatment Group (Experimental): RTC with Triple Antibiotic Study Drug
  Interventions: Drug: Experimental: Regeneration Treatment Group; Procedure: Control Non-Study Drug Group
- Control Non-study Drug Group (No Intervention): RTC on contralateral tooth with no study drug

INTERVENTIONS:
Drug: Experimental: Regeneration Treatment Group — Regenerative Root Canal Therapy using Triple Antibiotic Paste study drug
  Other Names: Regenerative RTC using Triple Antibiotic Paste study drug
  Arms: Regeneration Treatment Group
Procedure: Control Non-Study Drug Group — Endodontic RTC with no study drug
  Other Names: Root Canal Therapy
  Arms: Regeneration Treatment Group

SUMMARY:
The purpose of our study is to characterize the composition of the hard and soft tissues present after regenerative endodontic procedures in root canals of teeth previously diagnosed with the need for extraction for orthodontic treatment and incomplete root formation. Although the protocol addressed in this study is currently being used in clinical practice, there are no prospective clinical trials investigating its efficacy in stimulating continued root development and the nature of the newly formed tissues.

DETAILED DESCRIPTION:
Twenty subjects with permanent bilateral premolar teeth with incomplete root development and scheduled for extraction due to orthodontic requirement will be treated with a regeneration protocol. Teeth (n=20/group) will be extracted at 3 months following the regenerative protocol or the pulpectomy control. The protocol relies on disinfection of the canal space by copious irrigation with common endodontic irrigants and placement of a triple antibiotic paste (regenerative group) or calcium hydroxide dressing (control group) to disinfect the root for a period of one month. In each patient, both treatment arms will be performed. Thus, each treatment sample will have a contralateral matching control (paired designs). At the end of one month, the intracanal medicaments (triple antibiotic paste) is irrigated out of the canal and a blood clot is stimulated in the canal with the aid of endodontic files that are introduced into the periapical tissues; this blood clot will serve as a scaffold for tissue proliferation within the canal. The regenerative treatment tooth is then restored to prevent bacteria from the oral cavity from re-contaminating the canal space. For the contralateral control tooth, the medication will remain in the tooth until the extraction date. The subjects in this study will have the treated teeth extracted at 3 months after initial treatment. The extracted teeth from each study participant will be placed in storage medium until Immunohistochemical analysis with antibodies to characterize the tissue/cells within the canal.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria:

* Children ages 9-18 with bilateral premolars with incomplete root development scheduled for extraction for orthodontic reasons.
* Children who seem to be cooperative with dental treatment and able to indicate willingness to obtain treatment and participate in the study and who are capable of verbally expressing dissent.
* Parents who express understanding of study treatments and consent to treatment for their child of the regenerative procedure prior to the tooth extraction for orthodontic reasons .
* Healthy patients (ASA Class I or II physical status) with no systemic health problems that may interfere with healing and cell growth.

Tooth inclusion criteria:

* Permanent premolar teeth with immature root development and healthy pulps scheduled for extraction due to orthodontic requirements.
* Clinically confirmed teeth with good periodontal health assessed by periodontal probing depths of less than 4mm.

Exclusion Criteria:

Patient Exclusion Criteria:

* Parents and patients unable to give consent or express dissent.
* Patients who are unwilling to undergo the research and orthodontic dental treatment.
* Patients affected by tempromandibular joint disorders.
* Patients affected by known orofacial pain disorders.
* Patients with ASA Class III or IV physical status (Immuno-compromised patients including patients who self-report that they are an HIV carrier, undergoing steroid therapy or chemotherapy, or those who self-report with genetic or systemic diseases that could result in reduced immune response).

Tooth Exclusion Criteria:

* Teeth with vertical cracks that extend below the cemento-enamel junction.
* Teeth that cannot be isolated using a rubber dam.
* Teeth with non-odontogenic pathology.
* Teeth whose apices are fully developed, as determined radiographically and correlated with dental age of patient.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Histological identification of the mineralized tissue at the apical third of the root and the adherent cellular layer. | Following tooth extraction at the 3 month followup visit. Correlation of all data collected from the extracted teeth will occur at the completion of the study at year 5.
  Although we predict histological identification of dentin/odontoblasts (due to the proximity of the apical papilla and associated SCAP stem cells) using our scanning laser confocal microscopy system, our methods are sufficiently sensitive to permit identification of bone/osteoblasts and cementum/cementoblasts as alternative hypotheses.

SECONDARY OUTCOMES:
Whether stem cells enter the canal space when bleeding is stimulated through manipulation of the apical papilla. | Canal bleeding is evoked during the second treatment visit thirty days following the first treatment. Blood collected by paper points will be saved till the end of the study (year 5) for analysis.
  This secondary outcome measure will be conducted by measuring markers of stem cells prior to and after the formation of the blood clot. We predict that evoking bleeding into the root canal system will increase the delivery of mesenchymal stem cells.

CONTACTS AND LOCATIONS:
Overall Officials: Anibal R Diogenes, DDS, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Dubravko Pavlin, DMD, PhD, Principal Investigator — University of Texas Health Science Center San Antonio; Kenneth M Hargreaves, DDS, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States

REFERENCES:
- [Background] Thibodeau B. Case report: pulp revascularization of a necrotic, infected, immature, permanent tooth. Pediatr Dent. 2009 Mar-Apr;31(2):145-8. PMID 19455934